CLINICAL TRIAL: NCT00453180
Title: A Pilot Study of Oral N-Acetylcysteine in Children With Autism Spectrum Disorders
Brief Title: A Study of Oral N-Acetylcysteine in Children With Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Alliance for Autism Research (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0611-10
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive
Keywords: Autistic Disorder; Asperger's; PDD NOS; Pervasive Developmental Disorder; Autism; N-acetylcysteine; acetylcysteine; NAC; antioxidant; treatment; core symptoms; Autism Spectrum Disorders; Asperger's Disorder; Pervasive Developmental Disorder Not Otherwise Specified; Pervasive Developmental Disorders
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive; Autism Spectrum Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Target dose for n-acetylcysteine is 60 mg/kg/day. Capsules available in 300 mg and 600 mg strengths.
  Interventions: Drug: N-acetylcysteine
- 2 (Placebo Comparator): Subjects randomized to placebo arm will receive capsules identical in size and appearance to those subjects receiving study drug. Placebo capsules contain inactive ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Capsules available in 300 mg or 600mg strength. Target dose of n-acetylcysteine will be 60mg/kg/day TID. Dosage will be increased to this target dose from week 1 to week 3 barring side effects. Dose reduction will be allowed at any time for adverse side effects. Maximum dose of n-acetylcysteine will be 4200mg/day.
  Arms: 1
Drug: Placebo — Subjects randomized to placebo arm will receive placebo pill for duration of study.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether treatment with oral N-acetylcysteine (NAC) will improve behavior problems often associated with autism spectrum disorders.

DETAILED DESCRIPTION:
Autism is increasingly being recognized as a common disorder with enormous public health significance. The core symptoms of autism include severe deficits in social relatedness and communication, and interfering repetitive behavior. No medications have been shown to consistently improve any of these symptoms.

The central hypothesis of this study is that NAC will improve behavioral manifestations of autism which may include core or associated symptoms. We plan to test our hypothesis and complete the objectives of this project by pursuing the following specific aims:

* Evaluate the efficacy of oral NAC in a 12-week, double-blind, placebo-controlled study involving 32 children and adolescents with autism spectrum disorders.
* Evaluate the safety and tolerability of oral NAC in 32 children and adolescents with autism spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 12 years.
* Diagnosis of autistic disorder, Asperger's disorder, or PDD NOS.
* If taking concomitant psychotropic medications, the medication must be at a constant dose for 60 days with no dose changes planned for the duration of the trial.
* Able to swallow capsules.

Exclusion Criteria:

* Presence of any medical condition that significantly increases risk or hampers assessment (e.g., unstable hypertension or cardiac disease, unstable asthma, kidney disease, unstable seizure disorder, pregnancy or any other medical condition as determined by the investigator).
* Weight < 15 kg.
* Subjects taking concomitant medications or supplements known for their glutamatergic effects (e.g., dextromethorphan, D-cycloserine, amantadine, memantine, lamotrigine, riluzole) or antioxidant properties (high dose vitamin supplements, DMG, TMG, many alternative treatments) within 30 days of the baseline visit with the exception of short term use of dextromethorphan as needed as a cough suppressant. The use of this medicine must be stopped at least 7 days prior to the baseline visit. Regular multivitamins will be allowed.
* Subjects taking daily acetaminophen or nonsteroidal anti-inflammatory drugs within 30 days of the baseline visit.
* Profound mental retardation as evidenced by a mental age below 18 months.
* Subjects taking concomitant medications with the potential for pharmacokinetic or pharmacodynamic drug-drug interactions (e.g., carbamazepine) within 30 days of the baseline visit.
* Subjects who are likely to experience significant changes in their ongoing psychosocial or medical treatments for autism over the course of the trial (e.g., initiation of new behavioral therapy, initiation of new medication or alternative treatment [e.g., chelation]). Minor changes in ongoing treatment (e.g., missed therapy sessions due to holiday/vacation; planned break in therapy due to school holidays) will not be considered significant.
* History of prior treatment with NAC.
* Evidence of hypersensitivity/allergy to NAC.
* Presence of certain neurodevelopmental disorders such as Fragile X Syndrome, Tuberous Sclerosis, or other neurological disorders known to be associated with autism or autistic features.
* Diagnosis of Rett's disorder, childhood disintegrative disorder, schizophrenia, bipolar disorder, another psychotic disorder, or substance abuse disorder.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin H. Plawecki, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital, Riley Child and Adolescent Psychiatry Clinic, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Wink LK, Adams R, Wang Z, Klaunig JE, Plawecki MH, Posey DJ, McDougle CJ, Erickson CA. A randomized placebo-controlled pilot study of N-acetylcysteine in youth with autism spectrum disorder. Mol Autism. 2016 Apr 21;7:26. doi: 10.1186/s13229-016-0088-6. eCollection 2016. PMID 27103982
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Groups:
- N-acetylcysteine: Target dose for n-acetylcysteine is 60 mg/kg/day. Capsules available in 300 mg and 600 mg strengths.
  N-acetylcysteine: Capsules available in 300 mg or 600mg strength. Target dose of n-acetylcysteine will be 60mg/kg/day TID. Dosage will be increased to this target dose from week 1 to week 3 barring side effects. Dose reduction will be allowed at any time for adverse side effects. Maximum dose of n-acetylcysteine will be 4200mg/day.
- Placebo: Subjects randomized to placebo arm will receive capsules identical in size and appearance to those subjects receiving study drug. Placebo capsules contain inactive ingredients.
  Placebo: Subjects randomized to placebo arm will receive placebo pill for duration of study.
Period: Overall Study
Arm/Group | N-acetylcysteine | Placebo
Started | 16 | 15
Completed | 13 | 12
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 15 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.6 (2.5) | 8.2 (2.9) | 7.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Clinical Global Impression-Severity [Count of Participants; unit: Participants] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  Participants
    1. Normal, not al all ill | 0 | 0 | 0
    2. Borderline ill | 0 | 0 | 0
    3..Mildly ill | 0 | 0 | 0
    4. Moderatly ill | 6 | 9 | 15
    5. Markedly ill | 9 | 6 | 15
    6. Severly ill | 1 | 0 | 1
    7. Extremly ill | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression - Severity
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 12
Participants
  1.Normal, not at all ill | 0 | 0
  2.Borderline ill | 0 | 0
  3.Mildly ill | 3 | 0
  4.Moderately ill | 5 | 12
  5.Markedly ill | 5 | 0
  6.Severely ill | 0 | 0
  7.Extremely ill | 0 | 0

2. Primary Outcome: Clinical Global Impression - Improvement
Description: Clinical Global Impression - Improvement (CGI-I) is designed to take into account all factors to arrive at an assessment of response to treatment.
  The CGI-I scale ranges from 1 to 7 (1=very much improved; 2=much improved, 3=minimally Improved, 4=no change, 5=minimally worse, 6= much worse and 7=very much worse). Participants with a CGI-I score of 1 or 2 were classified as improved. Participants with a CGI score of 3, 4 or 5 were classified as no response. No participants scored 6 or 7.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 12
Participants
  Improved | 6 | 5
  No Response | 7 | 7

3. Secondary Outcome: Aberrant Behavior Checklist
Description: The Aberrant Behavior Checklist (ABC) is a 58-item measure of maladaptive behaviors and is used as a measure of drug effects. Each of the 58 items are rated from 0 (not at all) to 3 (severe).The ABC has 5 subscales: Irritability (15 items) ranging from 0 (not at all) to 45 (severe), Lethargy (16 items) ranging from 0 (not at all) to 48 (severe), Stereotypy (7 items) ranging from 0 (not at all) to 21 (severe), Hyperactivity (16 items) ranging from 0 (not at all) to 48 (severe), and Inappropriate Speech (4 items) ranging from 0 (not at all) to 12 (severe). Higher scores indicate a higher level of maladaptive behavior.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale
  Irritablity | 14.9 (14.0) | 12.0 (7.3)
  Lethargy | 10.0 (7.1) | 7.9 (4.7)
  Stereotypy | 3.9 (5.1) | 5.8 (4.0)
  Hyperactivity | 17.4 (16.4) | 15.1 (10.8)
  Inappropriate Speech | 4.1 (3.9) | 5.14 (3.5)

4. Secondary Outcome: Social Responsiveness Scale
Description: The Social Responsiveness Scale (SRS) is a 65-item scale that assesses social impairment in the aspects of social awareness, social cognition, social communication, social motivation and autistic mannerisms. Each item is scored from 0 (not true) to 3 (almost always true). The total SRS raw score may range from 0-195, where higher scores indicate greater severity.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 85.8 (34.9) | 89.1 (26.3)

5. Secondary Outcome: Pervasive Developmental Disorder Behavior Index
Description: The PDD Behavior Inventory (PDDBI) is a rating scale filled out by caregivers or teachers that was designed to assess children having a Pervasive Developmental Disorder (PDD; autism, Asperger disorder, PDD-NOS, or childhood disintegrative disorder). Both adaptive and maladaptive behaviors are assessed in the scale, making it useful for treatment studies in which decreases in maladaptive behaviors and improvements in adaptive social and language skills relevant to PDD are expected.
Time Frame: Week 12
Population: Less than 25% of participants in each group received a score on the PDDBI due to a significant floor effect. As a result, the data for these participants are not considered reliable given the significant floor effect.
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Vineland Adaptive Behavior Scales-II (VABS-II)
Description: The VABS-II is a semi-structured interview designed to assess adaptive functioning in the domains of communication, daily living skills and socialization. Items in each domain are rated as either 0 (does not), 1(sometimes) or 2(independently) performs a given behavior or skill. The communication domain has 99 items with scores ranging from 0-198. The daily living skills domain has 109 items with scores ranging from 0-218. The socialization domain has 99 items with scores ranging from 0-198. The domains scores are combined to form the adaptive composite score (ranging from 20-160). The raw scores from the communication, daily living skills and socialization domains along with the composite score were selected for use in this study. Higher scores indicate a higher level of adaptive functioning.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale
  Communication | 88.5 (32.5) | 95.0 (30.3)
  Daily Living Skills | 99.0 (37.1) | 98.6 (33.4)
  Socialization | 71.7 (18.7) | 75.9 (21.0)
  Adaptive Behavior Composite | 62.9 (17.1) | 60.5 (18.8)

ADVERSE EVENTS:
Time Frame: Twelve Weeks
Groups:
- Placebo: Subjects randomized to placebo arm will receive capsules identical in size and appearance to those subjects receiving study drug. Placebo capsules contain in active ingredients.
  Placebo: Subjects randomized to placebo arm will receive placebo pill for duration of study.
Arm/Group | N-acetylcysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 16/16 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine (N=16) | Placebo (N=15)
Aggression (Psychiatric disorders) | 3 | 2
Accidental arm injury (Musculoskeletal and connective tissue disorders) | 0 | 1
Appetite Increase (General disorders) | 1 | 0
Behavior Worse (Psychiatric disorders) | 1 | 2
Cold (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Difficulty Falling Asleep (Psychiatric disorders) | 4 | 1
Ear Infection (Ear and labyrinth disorders) | 2 | 1
Dry Mouth (General disorders) | 0 | 1
Elevated liver enzymes (Hepatobiliary disorders) | 1 | 0
Encopresis (Gastrointestinal disorders) | 0 | 1
Enuresis (Gastrointestinal disorders) | 1 | 1
Hand Movements (Nervous system disorders) | 0 | 2
Fever (General disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 3
Hives (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoglycemia (Endocrine disorders) | 1 | 0
Increased Swelling of Feet (Vascular disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Intermittent Dyspepsia (Gastrointestinal disorders) | 1 | 0
Itchy Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Nasal Cauterization (Surgical and medical procedures) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Poison Ivy (Skin and subcutaneous tissue disorders) | 0 | 1
Localized Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Scabies (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Picking/SIB (Psychiatric disorders) | 0 | 1
Stuttering (Nervous system disorders) | 1 | 0
Swollen neck lymph node of unknown origin (Endocrine disorders) | 1 | 0
Threats to hurt self (Psychiatric disorders) | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Weight Gain (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No